CLINICAL TRIAL: NCT03920189
Title: Left Diastolic Function in ARDS Mechanically Ventilated Patients
Brief Title: Echocardiographic Evaluation in ARDS Patients
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Davide Chiumello, Prof, University of Milan
Other Study IDs: ARDS-ECHO
Record Dates: First submitted 2019-04-16; First posted 2019-04-18 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Acute Respiratory Distress Syndrome; Mechanical Ventilation; Echocardiographic Ultrasound
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: echocariographic ultrasound — left ventricular diastolic function description

SUMMARY:
The purpose of this study is to assess the left diastolic function at different levels of in patients affected by the acute respiratory distress syndrome (ARDS)

DETAILED DESCRIPTION:
Introduction Left ventricular diastolic dysfunction (DD) is a clinical entity that remains poorly understood and identified in the intensive care unit (ICU) setting. In general, it is a syndrome defined by the presence of symptoms of congestive heart failure without sign of reduced left ventricle systolic dysfunction. Distinguishing diastolic heart failure from systolic heart failure is important because of differences in treatment and prognosis, even if often the two entities coexist, and some authors have proposed the hypothesis that diastolic LV dysfunction is essentially a precursor of systolic failure. At the base on DD there are multiple causes and multiple disorders. Among these, the impaired relaxation (common in ischemia and during systemic inflammatory states), an impaired peak left ventricular (LV) filling rate (with inadequate trans-mitral pressure gradient due to raised LV pressure or inability to generate negative LV pressure), the stiffness of LV (fibrosis and hypertrophy), and constriction (pericardial or compression from dilated right ventricle). Diastolic LV dysfunction is common in the ICU but often unrecognized. Its knowledge and determination of its severity may be useful to optimize circulatory support in critically ill patients. From this point of view, echocardiography is one of the most powerful diagnostic and monitoring tools available, providing the means to diagnose cardiac systolic or diastolic dysfunction, its underlying cause, and suggest therapeutic interventions. The aim of this study is to describe the presence and the grade of the eventually left diastolic dysfunction in ARDS patients and its possible correlation with the severity of illness and outcome.

Definitions and pathophysiology Diastolic heart failure is defined as a condition caused by increased resistance to the filling of one or both ventricles; this leads to symptoms of congestion from the inappropriate upward shift of the diastolic pressure-volume relation. Although this definition describes the principal pathophysiologic mechanism of diastolic heart failure, it is not clinically applicable. In a more practical definition diastolic heart failure is a condition that includes classic congestive heart failure findings with normal systolic function at rest, but with alteration in diastolic function. During DD the combination of active relaxation and passive myocardial compliance that normally maintain an adequate cardiac output are altered and left atrial pressure should be increased to maintain a satisfactory cardiac output. Different parameters have been used over the past two decades to describe the DD, so it is difficult to define its real incidence in critically ill patients. It seems to occur in about 30% of cases, and the majority of the studies tend to relate it with concomitant syndrome such as sepsis or clinical conditions such as respiratory weaning failure.

Left Diastolic dysfunction in ICU Most of the literature available investigated left DD in septic patient, and even if in the majority of these studies the patients were mechanically ventilated, only few information are available about the role of mechanical ventilation (MV) or the acute phase of lung injury.

With The advent of tissue Doppler imaging (TDI) has simplified echocardiographic estimation of ventricular relaxation and ventricular filling pressures, and the increasing number of studies in the field have showed that diastolic dysfunction is common in critically ill patients. The significance of diastolic dysfunction was recently highlighted by studies that demonstrated that TDI parameters might be prognostically useful in ICU population. More recent observations may help to clarify the scenario in these terms. An alteration in the E/e' ratio has been described in patients with septic shock and, although one study found that the E/e' ratio is an independent predictor of mortality [20], another investigation failed to find this association.

Left diastolic dysfunction in mechanical ventilated and ARDS patients It is well known that mechanical ventilation can induce hemodynamic compromise and that myocardial dysfunction and its consequences are not properly reflected by conventional hemodynamic parameters. Myocardial function can be assessed at the bedside using transthoracic echocardiography (TTE); however, the 2D echocardiographic measurements have been used to investigate predominantly the effects on systolic rather than diastolic ventricular function. Recently, TDI has provided more load-independent parameters to assess cardiac function, but its use is not widespread in ICU. For these reasons and probably because DD is greatly underestimated, there are few paper focused on mechanical ventilation and DD, most of them during weaning period, and almost none during the acute phase. What we know is that positive pressure ventilation can affect preload, afterload and ventricular compliance. The net effect in most situations is a decrease in cardiac output. However, the effect may be beneficial in the context of decompensated heart failure, where the decreased preload and afterload result in a return to a more productive part of the Starling curve.

More it is known in patients with prolonged weaning time. In this scenario, isolated diastolic dysfunction is present in about 22% up to 39% of patients. The increase in preload and afterload during MV may impair the LV compliance and determine a pulmonary edema. The fall in LV pressure during relaxation phase is a key determinant of diastolic function, and depends on intrinsic (contractility, LV stiffness) and extrinsic (preload, afterload) factors. Recently, has been suggested how the LV relaxation impairment with increased filling pressures may be a key mechanism of failed prolonged weaning trials. To summarize all these evidence, we could state that the elimination of positive ventilation increases LV preload and afterload and may induce some physiologic changes that can determine tachycardia and hypertension. Those are coincidentally two major determinants of diastolic dysfunction, as higher heart frequency reduces diastolic filling time and/or decreases coronary perfusion, and hypertension can exacerbate heart failure in patients with preserved ejection fraction. These findings suggest that echocardiography could be an excellent tool to guide the weaning process, helping to decide the best therapy to accomplish it.

Methods Consecutive mechanically ventilated patients will be enrolled within 48 hours after ICU admission with the diagnosis of ARDS. Demographic characteristics and respiratory mechanics variables (including esophageal pressure) will be recorded at two levels of positive end-expiratory pressure (PEEP); all patients will be study by a CT analysis at two levels of PEEP (5-45 cmh20) for the evaluation of recruitment potential, together with the computation of functional residual capacity (FRC). A well-trained cardiologist will perform a completed transthoracic echocardiography with the aim to describe the presence and the grade of left ventricular diastolic dysfunction (LVDD) applying a simplified definition of left DD, based on septal e', which is considered to be an index of myocardial relaxation, and the ratio of early diastolic velocity of mitral inflow to mitral annular velocity (E/e'), which has a strong association with left atrial pressure.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 or older and with a recent (<48h) diagnosis of ARDS, undergoing invasive mechanical ventilation

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive ARDS patients
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
echocardiographic ultrasound | day 1
  left ventricular dyastolic function

CONTACTS AND LOCATIONS:
Locations (1):
- ASST-Santi Paolo e Carlo, San Paolo Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No